CLINICAL TRIAL: NCT00567645
Title: Identification of the Role of Sympathetic Innervation in Heart Failure Patients Treated With Cardiac Resynchronization Therapy. A Pilot Study
Brief Title: Sympathetic Innervation of the Heart and Cardiac Resynchronization Therapy(CRT)
Acronym: PET-CRT
Status: Withdrawn | Type: Observational
Sponsor: University Medical Center Groningen (Other)
Responsible Party: Principal Investigator, I.C. Van Gelder, Prof.dr., University Medical Center Groningen
Other Study IDs: 16716
Record Dates: First submitted 2007-12-04; First posted 2007-12-05 (Estimated); Last update posted 2016-05-13 (Estimated); Status verified 2016-05

CONDITIONS: Sympathetic Innervation; Chronic Heart Failure

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to assess whether baseline sympathetic innervation in patients with chronic heart failure (CHF) is predictive for response to cardiac resynchronization therapy (CRT). And to assess whether response to CRT coincides with restoration of regional sympathetic innervation.

ELIGIBILITY:
Inclusion Criteria:

* Indication for CRT
* Stable optimal medication
* Non ischemic cardiomyopathy

Exclusion Criteria:

* Age less then 18 years
* Previous CRT
* Clinically relevant valvular heart disease or coronary artery disease
* Acute or chronic infection
* Untreated clinical hypo- or hyperthyroidism or < 3 months euthyroidism
* Uncontrolled hypertension, defined as a systolic blood pressure > 160 mm Hg and/or a diastolic blood pressure > 95 mm Hg
* A concurrent medical condition (i.e. alcohol or drug abuse or a severe progressive extra cardiac disease or M. Parkinson) or is unlikely to comply with the protocol
* Participation to a previous protocol involving radioactivity in the past year
* Pregnancy

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: chronic heart failure patients with CRT
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2007-07

PRIMARY OUTCOMES:
sympathetic innervation in patients with chronic heart failure (CHF) | 6 months

SECONDARY OUTCOMES:
NYHA class Echocardiographic parameters: LVEDD, LVESD, LVEF, LVESV,IVMD, and septal to lateral delay Hospitalization for heart failure Maximal oxygen consumption NT pro-BNP changes | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Isabelle C. Van Gelder, Prof, Principal Investigator — University Medical Center Groningen, departmen cardiology
Locations (1):
- University Medical Center Groningen, Groningen, Provincie Groningen, Netherlands